CLINICAL TRIAL: NCT03174314
Title: Feasibility and Efficacy of the VIS4ION Platform and Assistive Tactile and Auditory Communicating Devices in Low Vision Subjects
Brief Title: Feasibility and Efficacy of Assisstive Tactile and Auditory Communicating Devices
Acronym: VIS4ION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00317
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Visual Impairment
Keywords: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Visually impaired (Experimental): Visually impaired subjects will provide continuity across iterations of the testing, allowing for direct comparisons of responses within an individual for a single behavioral measure across different iterations of the device architecture and output configuration.
  Interventions: Behavioral: Standard object battery and training sequence
- Healthy controls (Active Comparator): Healthy (naive) subjects invaluable insights as well as a range of body types, cognitive abilities, and other idiosyncrasies that will keep our design and testing process from tailoring the device to a small set of individuals rather than the broader population.
  Interventions: Behavioral: Standard object battery and training sequence
- Thailand Site - Group A: Assistive Mode then Passive Mode (Experimental): During the first 15 days, group A will go through an assistive mode and then a passive mode for the next 15 days
  Interventions: Device: VIS4ION System
- Thailand Site - Group B: Passive Mode then Assistive Mode (Active Comparator): Group B will go through a passive mode for the first 15 days and then an assistive mode for the second half of the month
  Interventions: Device: VIS4ION System

INTERVENTIONS:
Behavioral: Standard object battery and training sequence — Used to examine human localization and identification performance. Object battery will include: trip hazards ('pucks' with various height/width combinations to represent children's toys, street debris, rocks, pets, etc.), furniture (chairs, desks, couches, benches), people, walls, and corridors. Objects will be recorded by placing them to the right or left on the path-of-travel. Raw sensor outputs for single obstacles and walls in isolation (trip-hazard pucks with 8 heights, chair, desk, person, wall) and the same set of single obstacles against a wall. This set of 23 raw sensor traces can be used in various combinations (e.g., encountering a curb and then a person, or a chair) to create a training sequence that will help experimentally naïve subjects to understand the correspondence between tactile stimulation and the real-world scenario it is intended to depict.
  Arms: Healthy controls; Visually impaired
Device: VIS4ION System — When in "Assistive Mode," participants will navigate campus while receiving navigation assistance (acquiring data and simultaneously providing assistance/audio feedback). When in "Passive Mode," participants will navigate campus wearing the backpack without receiving navigation assistant.
  Arms: Thailand Site - Group A: Assistive Mode then Passive Mode; Thailand Site - Group B: Passive Mode then Assistive Mode

SUMMARY:
This pilot study will integrate multi-sensor fusion techniques (software) to effectively combine information obtained from the newly embedded infrared, ultrasound, and stereo-camera-based sensor systems (hardware) that are implemented into the VIS4ION platform.

The core of this technology is based on 4 components: (1) a wearable vest with several distinct range and image sensors embedded. These sensors extract pertinent information about obstacles and the environment, which are conveyed to (2) a haptic interface (belt) that communicates this spatial information to the end-user in real-time via an intuitive, ergonomic and personalized vibrotactile re-display along the torso. (3) A smartphone serves as a connectivity gateway and coordinates the core components through WiFi, bluetooth, and/or 4G LTE, (4) a headset that contains both binaural, open-ear, bone conduction speakers (leaving the ear canal patent for ambient sounds) and a microphone for oral communication-based voice recognition during use of a virtual personal assistant (VPA).

Blindfolded-sighted, and blind subjects in a real-world, combined obstacle avoidance / navigation task will serve as an independent measure of overall improvements in the system as well as a roadmap for future avenues to enhance performance.

Further, a prospective, randomized crossover, controlled, non-blinded phase will be conducted in Thailand as part of this study to compare and evaluate effectiveness of the wearable vest for increasing navigation and quality of life.

DETAILED DESCRIPTION:
Investigators will try to develop algorithms that will recognize multiple objects and persons in real-time (enhanced scene interpretation for multi-object identification). And based on that, human-centered simulation trials and experiments for feasibility and efficacy of the platform's tactile and auditory 'communication' outputs will be conducted. Finally auditory and tactile 'prompts' (system output) based on the end user's immediate needs based on initial testing results, will be integrated into the platform.

Additional activities will occur at the Thailand site. In the second phase, an improved system will be tested in an extended-use experiment, detecting for health-related changes in our participants (increased mobility and QoL). The study team will further test the generalizability of the new mapping technology in a more challenging environment, testing system performance using metrics, comparing results between current and previous systems.

ELIGIBILITY:
Inclusion Criteria:

* People with visual impairments of all different levels and etiologies.

Exclusion Criteria:

* Significant cognitive dysfunction (score <24 on Folsteins' Mini Mental Status Examination)
* Previous neurological illness, complicated medical condition;
* Significant mobility restrictions; people using walkers and wheelchairs
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Correct Responses by Feedback Devices | Month 6
  Assessment of ability of the feedback devices (vibrating belt- wrist band/haptic interface and audio output/open-ear headset) to provide correct responses on alternative force choice tasks during simulation experiments.
Total Time to Complete Activities of Daily Living | Month 6
  Such activities can include navigation, shopping and cooking.
Path Length | Month 6
  Total length of the path taken when participants perform navigation task.
Success Rate | Month 6
  Percentage of participants who achieve the destination and/or target in the navigation task.

SECONDARY OUTCOMES:
Change in International Physical Activity Questionnaire (IPAQ) Score | Baseline, Month 6
  7-item questionnaire assessing the types and intensity of physical activity and sitting time that people do as part of their daily lives; the total score is total physical activity, which is quantified in metabolic equivalent (MET) minutes per week.
Change in World Health Organization Quality of Life (WHOQOL)-BREF Score | Baseline, Month 6
  WHOQOL-BREF is a 26-item questionnaire assessing how patients have felt about their quality of life and health over the past 4 weeks. Each item is rated on a scale from 1-5. The raw score is the sum of responses and is rescaled to a total score of 0-100; higher scores indicate greater health states.
Change in Visual Functioning Questionnaire - 25 (VFQ-25) Score | Baseline, Month 6
  25-item assessment of how participants feel about their vision or vision condition. Each item is rated on a scale from 1-6. The raw score is the sum of responses and is converted to a 0-100 scale for the total score; higher scores indicate greater visual functioning.

CONTACTS AND LOCATIONS:
Overall Officials: John R Rizzo, MD, Principal Investigator — NYU Langone Health
Locations (4):
- New York University School of Medicine, New York, New York, United States
- Thailand (3):
  - Mahidol University College of Music, Engineering, Science, Religious Studies, Social Sciences and Humanities, Salaya
  - Mahidol University International College, Salaya
  - Ratchasuda College, Mahidol University, Salaya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beheshti M, Naeimi T, Hudson TE, Feng C, Mongkolwat P, Riewpaiboon W, Seiple W, Vedanthan R, Rizzo JR. A Smart Service System for Spatial Intelligence and Onboard Navigation for Individuals with Visual Impairment (VIS4ION Thailand): study protocol of a randomized controlled trial of visually impaired students at the Ratchasuda College, Thailand. Trials. 2023 Mar 7;24(1):169. doi: 10.1186/s13063-023-07173-8. PMID 36879333